CLINICAL TRIAL: NCT06346860
Title: Comparing Postoperative Analgesic Effects of Intrathecal Morphine With Modified Thoracoabdominal Nerve Block Through Perichondral Approach in Major Abdominal Surgery
Brief Title: Comparing Intrathecal Morphine With Modified Thoracoabdominal Nerve Block Through Perichondral Approach in Major Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Beliz Bilgili, Associate Professor, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 09.2024.241
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Opioid Use; Postoperative Pain
Keywords: intrathecal morphine; Modified Thoracoabdominal Nerve Block Through Perichondral Approach
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Thoracoabdominal Nerve BlockThrough Perichondral Approach and PCA (Active Comparator): Modified Thoracoabdominal Nerve BlockThrough Perichondral Approach and Intravenous Patient Controlled Analgesia
  Interventions: Procedure: Regional Block Comparison
- Intrathecal Morphine and Intravenous Patient Controlled Analgesia (Placebo Comparator): Intrathecal Morphine 200 mcg and Intravenous Patient Controlled Analgesia (1 mg/ml morphine, 1 cc bolus, 7 min. locked
  Interventions: Procedure: Regional Block Comparison

INTERVENTIONS:
Procedure: Regional Block Comparison — Comparing postoperative pain and opioid consumption in groups

SUMMARY:
Abdominal surgery causes severe postoperative pain due to retraction of the abdominal wall and direct manipulation of visceral organs. It leads to delayed postoperative recovery, increased postoperative morbidity and mortality. Intrathecal morphine, epidural analgesia and patient-controlled intravenous analgesia are used in postoperative pain management of abdominal surgeries. Intrathecal morphine is frequently used in many centers because it provides effective pain control. However; morphine has undesirable effects such as urinary retention, postoperative nausea and vomiting, and respiratory depression. Modified thoracoabdominal nerves block through perichondrial approach is a technique defined by the modification of the thoracoabdominal nerves block through perichondrial approach, in which local anesthetics are delivered only to the underside of the perichondral surface. The primary implication of this study is to compare postoperative pain scores and opioid consumption in patients undergoing major abdominal surgery with intrathecal morphine or modified thoracoabdominal nerves block through perichondrial approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Patients undergoing major abdominal surgery

Exclusion Criteria:

* Patients with solid organ dysfunction
* Patients who receive opioid or corticosteroid medication prior to surgery
* Patients with bleeding diathesis
* Patients with psychiatric disorders
* Patients who can not be contacted after surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Comparison of postoperative opioid consumption between two groups via Patient Controlled Analgesia (PCA) device | 48 hours
  Intravenous patient-controlled analgesia (PCA) is a system of opioid delivery that consists of an infusion pump interfaced with a timing device. Intravenous morphine consumption will be recorded via PCA device, then it will be documented in mg/kg units.

SECONDARY OUTCOMES:
Postoperative pain assessment with Numeric Rating Scale (NRS) | 48 hours
  In a Numerical Rating Scale (NRS), patients are asked to choose the number
Comparison of the frequency of treatment related complications | 48 hours
  Bradycardia, hypotension, sedation, respiratory depression, urinary retention, itching, need for rescue analgesics.
Participant satisfaction | 48 hours
  Whether the patient is very pleased/ satisfied/ unsatisfied/ complainant with the pain treatment will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided